CLINICAL TRIAL: NCT05272488
Title: A Combined Treatment of Manual Therapy and Nervous Vagus Stimulation Versus a Treatment of Manual Therapy Isolated in Patients With Myogenic Temporomandibular Disorders
Brief Title: A Combined Treatment of Manual Therapy and Nervous Vagus Stimulation in Patients With Myogenic Temporomandibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIM/2021/6/144
Record Dates: First submitted 2021-11-17; First posted 2022-03-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Temporomandibular Joint Disorders; Pain
Keywords: Temporomandibular Joint; Manual therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Musculoskeletal Manipulations; Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy and nervous vagus stimulation (Experimental): Subjects will received manual therapy combined with nerve vagus stimulation.
  Interventions: Other: Manual therapy and vagus nerve stimulation
- Manual therapy (Active Comparator): Subjects will received isolated manual therapy techniques.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy and vagus nerve stimulation — A neurodinamic intervention of vagus nerve through deep breaths involving diaphragm muscle and manual therapy techniques.
  Arms: Manual therapy and nervous vagus stimulation
Other: Manual therapy — Manual therapy techniques. Joint manipulation techniques for temporomandibular joints and Soft tissue techniques for the muscles
  Arms: Manual therapy

SUMMARY:
Temporomandibular disorders (TMD) are one of the most important Public Health issues in the world and its incidence has increased over the years. The Physiotherapy and manual therapy techniques has shown its efficacy to reduce pain and to improve jaw functionality in patients with TMD. Until now, treatment targets has been the muscle and joint, but clinicians has not taken into account the innervation and how the nerve can have an influence in pain or jaw functionality.

In this sense, it is known that there is a relationship between jaw innervation and vagus nerve, a parasympathetic nerve which is easily stimulable, due to its connection with the respiratory system, taking deep breaths using the diaphragm.

Therefore, our hypothesis is that a treatment in which clinicians combine manual therapy and nerve vagus stimulation could have better effects (reducing pain, increasing range of motion in temporomandibular joints and improving quality of life in patients with TMD) than a isolated manual therapy treatment.

With this purpose will be selected 20 subjects to participate in our study divided in two groups. Both groups will received 4 sessions of physiotherapy (one each 7 days during one month) and also will be thought to do own treatment those days the subjects does not come to the clinic until the study will have finished (the interventional period last two months). Both groups will received the same manual therapy techniques but only the experimental group will be treated with nerve vagus stimulation technique.

One member of the group who will not participated in the interventions will be in charge of do evaluations (1 each month/ a total of 3 evaluations) following different questionaries to assess the primary variables of the study: chronic pain level, jaw functionality, physical symptoms level, range of motion and distress level.

DETAILED DESCRIPTION:
The aim of the study is to check whether vagus nerve stimulation (VNS) combined with manual therapy (TM), given its neuroanatomical relationship with the structures involved in pain in the TMJ, is more effective in reducing pain, increasing joint range and increasing the quality ofthe patient lives than TM alone.

The research team is made up of three physiotherapists. It has been decided to distribute the tasks as follows:

* Physiotherapist 1 will be in charge of the treatment of all patients.
* Physiotherapist 2 will be responsible for screening the sample and evaluating the study.
* Physiotherapist 3 will be in charge of analyzing the results and statistics. This component of the team, being blinded and not knowing the group of origin of the patient, will be able to interpret the results without any type of convenience bias, showing absolutely transparency in the elaboration of the conclusions.

Once the screening will be completed, the patients will be divided into two groups: an experimental group (TM + ENV) and a control group (TM + ENV placebo).The randomization will be carried out through the statistical program Epidat 4,237 9 obtaining two homogeneous groups. Each patient will be assigned a code with the aim that the physiotherapist who is in charge of the statistical analysis is not able to establish links between the data and the subjects to which it refers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of myogenic pain according to the CD / TTM diagnostic criteria.
* Presence of pain during the last 30 days.
* Patients with decreased jaw function and mobility due to pain.
* Patients who have not received physiotherapy treatment in the last 3 weeks.
* Patients of legal age.

Exclusion Criteria:

* Patients with drug treatment: sedatives, anti-inflammatories, antidepressants, anxiolytics or muscle relaxants.
* Patients with cardiac pacemakers and implanted defibrillators. Patients diagnosed with severe cardiorespiratory and / or respiratory diseases, carcinogenic processes, infectious processes and / or systemic pathologies.
* Clinical diagnosis of temporomandibular disorder of joint or mixed origin according to the Diagnostic Criteria for Temporomandibular Disorders (CD / TMD).
* Patients with psychiatric or psychological disorders, intellectual or motor deficiencies that, due to their nature, prevent them from correctly performing the prescribed exercises, correctly following the physiotherapist's instructions or understanding the questionnaires and / or measurement scales of the variables.
* Patients with dental processes scheduled during the study period or who have undergone surgery in the last 3 months.
* Patients with suspicion or certainty that their pain has appeared as a consequence of a local or general trauma.
* Patients diagnosed with fibromyalgia, neuropathic pain or degenerative diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Patient´s state of health | Change from baseline at 2 months
  An interpretation of the improvement of patient´s state of health related with temporomandibular disorders taking into account other improvements in differents areas/variables which will be described as secondary outcomes
Graded Chronic Pain Scale (CPGS) | Change from baseline at 2 months
  The CPGS is a multidimensional measure that assesses 2 dimensions of overall chronic pain severity: pain intensity and pain-related disability. It is suitable for use in all chronic pain conditions.The 3 subscale scores (characteristic pain intensity, disability score, and the disability points score) are used to classify subjects into 1 of the 5 pain severity grades: grade 0 for no pain, grade I for low disability-low intensity, grade II for low disability-high intensity, grade III for high disability-moderately limiting, and grade IV for high disability-severely limiting.

SECONDARY OUTCOMES:
Range of motion (Opening without pain, Maximum Opening, Lateral movements and Protrusion movement) | Change from baseline at 2 months
  All of them were measured in millimeters using a rule. The evaluator take 3 measures of each movement and the final outcome was the average of these 3 measures.
Jaw Functional Limitation Scale | Change from baseline at 2 months
  The JFLS-20 is a scale that assesses the limitation of jaw function during chewing, mobility, and verbal and non-verbal communication.The maximum score is 20. Lower scores denote lower aw functional limitation and higher scores denote higher jaw functional limitation.
The Patient Health Questionnaire (PHQ-15) | Change from baseline at 2 months
  The PHQ-15 is comprised of 15 items and assesses non-specific physical symptoms, also referred to as functional symptoms or medically unexplained symptoms.PHQ-15 scores of 5, 10, 15, represented cutoff points for low, medium, and high somatic symptom severity, respectively
Distress Level PHQ-4 | Change from baseline at 2 months
  This one was assesed using PHQ-4. The PHQ-4 is comprised of two 2-item subscales, anxiety and depression, and it is intended to be an ultrabrief screener for distress as the composite construct of anxiety and depression.Total scores range from 0 to 12, with higher scores indicating greater psychological distress

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Ferragut-Garcías, PhD, Study Chair — Universidad Islas Baleares
Locations (3):
- Spain (3):
  - Clinical University Physiotherapy and pain, Alcalá de Henares, Madrid
  - Martinez-Merinero, Patricia, Alcalá de Henares, Madrid
  - Physioterapy and Pain center research, Alcalá de Henares, Madrid